CLINICAL TRIAL: NCT04813861
Title: Sequential Treatment of Hepatocellular Carcinoma by Transarterial Chemoembolization and Local Ablation or External Radiation
Acronym: CELPerCutCHC
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Valérie LAURENT, MD, PhD, Central Hospital, Nancy, France
Other Study IDs: 2020-PI199-99
Record Dates: First submitted 2021-03-21; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Transarterial Chemoembolization; Stereotactic body radiotherapy; Radiofrequency Ablation; Microwave Ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatocellular carcinoma (HCC) can present itself in many forms (size, number of lesions) for the treatment of which a therapeutic panel can be elaborated and layered. If a curative treatment cannot be considered in case of an HCC classified in an intermediate stage, a Transcatheter Arterial Chemoembolization (TACE) can be proposed. In case of a partial response or the treatment of some lesions of a multifocal HCC, a combined treatment by stereotaxic radiotherapy (CK), radiofrequency ablation (RFA) or microwave ablation (MWA) may be initiated in accordance with a decision of the multidisciplinary consultation meeting.

The aim of this study was to evaluate the clinical outcome of HCC receiving MWA, RFA or CK after downstaging with TACE.

ELIGIBILITY:
Inclusion Criteria:

* a HCC treated by TACE followed by RFA, MWA and/or CK
* from 01/2010 to 12/2020
* treated by Nancy Regional University Hospital (TACE, RFA, MWA) and Institut de Cancérologie de Lorraine (CK)

Exclusion Criteria:

* Combined treatment over one year following the last TACE
* No baseline, in between or after combined treatment imaging
* Lesion appeared after TACE treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been treated for HCC by TACE, followed by additional treatment with RFA, MWA or CK in the following year, between January 2010 and December 2020 by Nancy Regional University Hospital (TACE, RFA, MWA) and Lorraine Institute of Cancer (CK)
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2010-01-04 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Lesion Response | 4-6 weeks after BWA or RFA or 3-6 months after CK
  Lesion response after combined treatment

SECONDARY OUTCOMES:
Delayed Lesion Response | 1 year after BWA, RFA or CK
  Lesion response a year after combined treatment

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Nancy, France